CLINICAL TRIAL: NCT03446391
Title: Matched Pair Study to Assess Influence of Kinematic Versus Mechanical Alignment in Total Knee Replacement
Brief Title: Matched Pair Study - Kinematic Vs Mechanical Alignment
Status: Completed | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P02.010.18
Record Dates: First submitted 2018-02-19; First posted 2018-02-26 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee; Joint Disease
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Kinematic alignment with GMK Sphere®: Patients enrolled prospectively with surgeries planned to get kinematic alignment
  Interventions: Procedure: Kinematic alignment; Device: GMK Sphere®
- Mechanical alignment with GMK Sphere®: Historical group who had mechanical alignment, match-paired with the prospective group
  Interventions: Procedure: Mechanical alignment; Device: GMK Sphere®

INTERVENTIONS:
Procedure: Kinematic alignment — The principle for kinematically aligning the femoral component is to remove the correct amount of bone and cartilage from the distal and posterior femur after accounting for wear and saw blade kerf, so that the total thickness of the missing and removed tissue matches the thickness of the femoral component.
  Groups: Kinematic alignment with GMK Sphere®
Procedure: Mechanical alignment — Classic mechanical alignment (MA) in total knee arthroplasty (TKA) is meant to co-align the prosthetic components to the mechanical axes of the femur and tibia and restore neutral overall limb alignment
  Groups: Mechanical alignment with GMK Sphere®
Device: GMK Sphere® — The GMK Sphere® is a total knee prosthesis . The design of the GMK Sphere® is characterized by a spherical medial femoral condyle and an asymmetrical fixed tibial UHMWPE polyethylene insert with a concave spherical medial compartment.

SUMMARY:
The aim of this study is to evaluate postoperative knee function after total knee arthroplasty performed according to the anatomical alignment and compare these results to those of a matched historical cohort of patients operated with mechanical alignment.

DETAILED DESCRIPTION:
The 25 patients, of the Kinematic group, are prospectively enrolled. While, the data of patients of the Mechanical group, are retrospectively collected from an historical collection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with disease that meets the indications for use for Medacta implants defined by this study (on-label use).
2. Patients necessitating primary Total Knee Replacement
3. Patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to the patient's surgery.

Exclusion Criteria:

1. Those with one or more medical conditions identified as a contraindication defined by the labeling on Medacta implants used in this study.
2. Previous osteotomy around the knee
3. Ligament instability likely to require higher level of constraint
4. Previous infection or inflammatory disease
5. Extraarticular deformities for which a femoral intramedullary guide rod can't be inserted into the canal and use of Computer Assisted Orthopaedic Surgery (CAOS) or Patient Specific Instrumentation (PSI) is required.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited during the preoperative visit at the investigational site. All patients scheduled for a total knee replacements, meeting the inclusion criteria and none of the exclusion criteria will be invited to the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Compare clinical outcomes of mechanical vs kinematic with new Knee Society Score | 1-year follow-up
  The new KSS (from the publication of 2011, Giles R. Scuderi MD "The New Knee Society Knee Scoring System" Clin Orthop Relat Res (2012) 470:3-19) includes a part filled by the surgeon and one by the patient. The first outcome is focused on the "Functional Activities" subscore, excluding the "Discretionary knee activities". The maximum is 85 points while the minimum is -10 points. The "Functional Activities" score includes 3 subscores: WALKING AND STANDING (min -10, max 30), STANDARD ACTIVITIES (min 0, max 30) and ADVANCED ACTIVITIES (min 0, max 25)

SECONDARY OUTCOMES:
Patient functional improvement, satisfaction and symptoms | 1-year follow-up
  The functional improvement, satisfaction and symptoms is the sum of the following subscores of the new KSS: "Functional Activities", "Patient Satisfaction" and "Symptoms"
Residual deformity | 1-year follow-up
  The residual deformity is evaluated by long axis Xray analysis: HKA angle
Flexion-extension contracture | 1-year follow-up
  The flexion-extension contracture is evaluated by a subscore of the new KSS: "Joint motion"
Self-reported pain, function and stiffness | 1-year follow-up
  These aspects are evaluated through KOOS score
Ability to forget about artificial joint | 1-year follow-up
  Through the use of the Forgotten Joint Score

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vinzenz Krankenhaus Brakel, Brakel, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided